CLINICAL TRIAL: NCT05602103
Title: Identification of Anticancer Drugs Associated With Cancer Therapy-related Cardiac Dysfunction Reporting in Pediatrics - Analysis of the WHO Pharmacovigilance Database
Brief Title: Cancer Therapy-related Cardiac Dysfunction Occuring in Children Treated by Anticancer Drugs for Malignancies
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco_112022
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-04

CONDITIONS: Malignancies; Cardiovascular Diseases; Children, Only
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: use of anticancer drugs in monotherapy or in combination therapy — Cases of cancer therapy-related cardiac dysfunction associated with anticancer drugs will be identify and describe

SUMMARY:
Little is known about cancer therapy-related cardiac dysfunction occuring in children treated by anticancer drugs for malignancies. Here the investigators use VigiBase (http://www.vigiaccess.org/), the World Health Organization (WHO) database of individual safety case reports, to identify and describe cases of cancer therapy-related cardiac dysfunction associated with anticancer drugs.

ELIGIBILITY:
Inclusion Criteria:

* cases reported in the World Health Organization (WHO) database of individual safety case reports (vigibase)
* related to children
* and reported, or not, cancer therapy-related cardiac dysfunction

Exclusion Criteria:

* cases reported in the World Health Organization (WHO) database of individual safety case reports (vigibase) related to adult patients

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cases reported in the World Health Organization (WHO) database of individual safety case reports (vigibase) related to children and reported, or not, cancer therapy-related cardiac dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-11-05 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-06 (Estimated)

PRIMARY OUTCOMES:
cancer therapy-related cardiac dysfunction associated with anticancer drugs | from inception to the April 31, 2024
  identification and description of cases of cancer therapy-related cardiac dysfunction associated with anticancer drugs in the World Health Organization (WHO) database of individual safety case reports (vigibase)

SECONDARY OUTCOMES:
Association between cancer therapy-related cardiac dysfunction and anticancer drug exposure in the World Health Organization (WHO) database of individual safety case reports (vigibase) | from inception to the April 31, 2024
  Disproportionnality analyses in Vigibase (IC025 and/or ROR) perfomed on cases reported in the World Health Organization (WHO) database of individual safety case reports (vigibase)
Description of the malignancies for which the incriminated drugs have been prescribed | from inception to the April 31, 2024
  Cases reported in the World Health Organization (WHO) database of individual safety case reports (vigibase)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Alexandre, MD, PhD, Principal Investigator — Caen Normandy University Hospital, France

IPD SHARING:
Plan to Share IPD: No